CLINICAL TRIAL: NCT07329777
Title: Atropine in the Treatment of Myopia Study in Malaysia (ATOM-MY): A Randomized, Double-Blind Study to Demonstrate the Efficacy and Safety of Eye Drop Formulations (Atropine Sulphate 0.025 % w/v Eye Drops vs Placebo) in the Management of Controlling Progression of Myopia in Children.
Brief Title: Atropine in the Treatment of Myopia Study in Malaysia
Acronym: ATOM-MY
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: IDB VisionCare SDN BHD (Industry)
Collaborators: Singapore National Eye Centre (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CT01-ATOM-MY-2022
Record Dates: First submitted 2025-09-16; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Myopia Progression

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Atropine Sulphate 0.025% w/v Eye Drops (Active Comparator): Participants will be instructed to administer one drop of Atropine Sulphate 0.025% w/v Eye Drops into each eye once daily at bedtime for a duration of 24 months.
  Interventions: Drug: Low dose atropine sulfate eye drops
- Placebo (Placebo Comparator): Participants will be instructed to administer one drop of Placebo Eye Drops into each eye once daily at bedtime for a duration of 12 months and Atropine Sulphate 0.025% w/v Eye Drops from 13-24 months onwards.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Low dose atropine sulfate eye drops — Atropine Sulphate 0.025% w/v Eye Drops
  Arms: Atropine Sulphate 0.025% w/v Eye Drops
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This clinical trial is designed to assess the efficacy and safety of Atropine Sulphate 0.025% w/v Eye Drops compared to placebo in a randomized, double-blind, placebo-controlled study for the management of myopia progression in children.

DETAILED DESCRIPTION:
Myopia represents the most prevalent refractive error globally, with its incidence rising significantly over recent decades, particularly in East Asian populations. Current projections estimate that by the year 2050, nearly 50% of the global population will be affected by myopia, with approximately 10% classified as high myopes. High myopia is characterized by axial elongation of the eye and is associated with an elevated risk of severe ocular complications, including early-onset cataracts, glaucoma, retinal detachment, choroidal neovascularization, myopic macular degeneration, and macular hemorrhage. Given its increasing prevalence and potential for vision-threatening outcomes, myopia constitutes a substantial public health issue, contributing to considerable healthcare and socioeconomic burdens. Therefore, the development of safe and effective interventions to mitigate the progression of myopia is of critical importance.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female children between 5 to 10 years of age.
2. Children with refractive error of spherical equivalent -1.00 D up to -6.00 D in each eye.
3. Children with active myopia progression of at least spherical equivalent -0.50 D within the last 12 months.
4. Children with astigmatism of less than -1.50 D
5. Children having distance vision correctable to logMAR 0.2 or better in both eyes.
6. A difference between non-cycloplegic subjective spherical refraction and cycloplegic subjective spherical refraction of not greater than -1.00 D.
7. Children with normal intraocular pressure of not greater than 21 mmHg in either eye.
8. Children with normal ocular health other than myopia.
9. Children must be in good general health with no history of cardiac or respiratory diseases as per investigator's discretion and does not affect the study treatment or subsequent follow-ups.
10. No asthma-requiring medications in the past one year.
11. No known allergy to atropine, cyclopentolate, proparacaine and benzalkonium chloride.
12. Willing and able to comply with scheduled visits and other study procedures.
13. Written Informed Consent from parent and assent from child has been obtained.

Exclusion Criteria:

1. History of hypersensitivity or allergy to study drug and/or any of the study medication ingredients.
2. Children with prior and/or concomitant use of other myopia control drugs, contact lens or spectacles (except normal spectacles including tinted/anti-glare glasses) etc.
3. Children with congenital myopia.
4. Children using Ortho K and Myopia Lens.
5. Children with ocular or systemic diseases which may affect vision or refractive error.
6. Children with any ocular condition wherein topical atropine is contraindicated.
7. Children with defective binocular function or stereopsis.
8. Children with amblyopia (lazy eyes) or manifest strabismus including intermittent tropia.
9. Previous or current use of atropine or pirenzepine.
10. Children with any other conditions precluding adherence to the protocol including unwillingness to refrain from the use of other myopia control drug, contact lens or spectacles (except normal) spectacles including tinted/anti-glare glasses) etc. for the duration of the study.
11. Children with any other condition which may put the subject to risk during study or affect study results based on investigator's judgement.
12. Children participated in any clinical study within 30 days prior to randomization.

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 144 (Estimated)
Dates: Start 2025-09-17 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2029-09 (Estimated)

PRIMARY OUTCOMES:
To demonstrate the superiority of eye drop formulation (Atropine Sulphate 0.025% w/v Eye Drops) against placebo determined by Spherical equivalent | 12 months
  Spherical equivalent refraction determined by cycloplegic autorefraction from baseline to 12 months at each visit.

SECONDARY OUTCOMES:
To demonstrate continued efficacy of eye drop formulation (Atropine Sulphate 0.025% w/v Eye Drops) of 24 months with the comparison of 12 months by spherical equivalent | 24 months
  Determination of rate of progression in year 2 vs year 1 via Spherical equivalent refraction as determined by cycloplegic autorefraction of 24 months with the comparison of 12 months.
To demonstrate the superiority of eye drop formulation (Atropine Sulpahte 0.025% w/v Eye Drops) against placebo by axial length | 12 months
  Axial length as determined by non-contact partial coherence interferometry from baseline to 12 months at each visit.

CONTACTS AND LOCATIONS:
Locations (2):
- Malaysia (2):
  - Hospital Pakar Kanak-Kanak UKM, Kuala Lumpur, Cheras
  - Universiti Malaya Medical Centre, Kuala Lumpur, Petaling Jaya

IPD SHARING:
Plan to Share IPD: Undecided